CLINICAL TRIAL: NCT04456114
Title: Micro-abrasive Blasting vs Acid Etching of Orthodontic Bracket Bases: A Scanning Electron Microscope Study and an Eighteen Month Randomized Clinical Control
Brief Title: Micro-abrasive Blasting vs Acid Etching of Orthodontic Bracket Bases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Owais Khalid Durrani, Professor of Orthodonitcs, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIDC/IRB/06/06/2020
Record Dates: First submitted 2020-06-27; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Orthodontic Appliances

STUDY DESIGN:
Intervention Model Description: parallel-group, split mouth, triple blinded, randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acid etched brackets (Experimental): Stainless steel bracket base etched with 10% Hydrofluoric acid for 1 minute
  Interventions: Device: Acid etched brackets
- Sandblasted brackets (Active Comparator): Stainless steel bracket sandblasted base
  Interventions: Device: Sandblasted brackets

INTERVENTIONS:
Device: Acid etched brackets — The brackets will be bonded to the teeth with composite on the same patient in a split mouth design and observed for bracket debonding for 18 months
  Arms: Acid etched brackets
Device: Sandblasted brackets — The brackets will be bonded to the teeth with composite on the same patient in a split mouth design and observed for bracket debonding for 18 months
  Arms: Sandblasted brackets

SUMMARY:
To describe a method of acid etching the base of a bracket, and to compare the bond failures between micro-abrasive blasted (sandblasted) brackets and acid etched brackets over an eighteen month period

DETAILED DESCRIPTION:
The aims of this randomized control trial are:

1. To describe a method to chemically etch the bases of stainless steel orthodontic brackets.
2. To observe the changes in the micro-structure of the brackets with sandblasted bases and acid-etched bases under an electron microscope.
3. To compare the failure of orthodontic brackets with a chemical etched base versus a sandblasted base bonded with composite using the conventional acid etch technique, over a follow-up of 18 months

ELIGIBILITY:
Inclusion Criteria:

* Patients about to undergo fixed orthodontic therapy

Exclusion Criteria:

* Patients with cavities, history of fixed orthodontic therapy, recent bleaching

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Bond Failure Rate | 18 months after placement of brackets on the teeth
  To compare the bond failure rates between acid etched and sandblasted brackets. Done by calculating and comparing the percentages of bracket breakages between the acid etched and sandblasted bracket quadrants.

CONTACTS AND LOCATIONS:
Overall Officials: Owais K Durrani, FFDRCSI, Principal Investigator — Riphah International University
Locations (1):
- Islamic International Dental College, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No